CLINICAL TRIAL: NCT00966862
Title: The Glycemic Effect of Taking a Supplementation of Orange Juice With Fibers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC-09-NV-237-CTIL
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-05

CONDITIONS: Healthy People

INTERVENTIONS:
Other: Other: Dietary Fibers

SUMMARY:
The aim of this study is to investigate the glycemic effect of supplementation Fibers in orange juice.

This will be a double-blind parallel controlled study. Each subject will serve as his own control.

Study population will include 10 subjects. The subjects will be randomly assigned to receive one of two juices in occasion, in two visits. Each drink will be containing orange juice with\without fibers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Age 60 >18 years
* Written informed consent
* Consumers of orange drinks: freshly squeezed juices, commercial pasteurized juices and / or orange soft drinks
* Regular eating pattern

Exclusion Criteria:

* Patients with chronic disease sach as:

  * diabetes,
  * cancer,
  * C.O.P.D.,
  * metabolic syndrome,
  * overweight,
  * kidney failure,
  * heart disease,
  * osteoporosis.
* Antibiotic treatment in the last 4 weeks
* Subjects on regular probiotic or prebiotic supplementation, unless they do 2 weeks of wash out.
* Subjects with intestinal disorders such as: IBD, IBS, celiac, colon cancer.
* Subjects after intestinal surgery.
* Use of medicines for lowering cholesterol (simvastatin), sugar control
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2009-09; Primary Completion 2010-02 (Estimated); Study Completion 2010-05

PRIMARY OUTCOMES:
To investigate the Glycemic Effect by drawing blood for glucose and insulin

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof', Principal Investigator — Suorasky Medical Center
Locations (1):
- Suorasky Medical Center, Tel Aviv, Israel